CLINICAL TRIAL: NCT03851458
Title: Consumption of More Ideal Food Options (COMIDA: Consumo de Opciones Más Ideales De Alimentos)
Acronym: COMIDA
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Make the Road New York (MRNY) (Unknown); Mexican Coalition for the Empowerment of Youth and Families (Unknown); The City College of New York (Other); Mexican Consulate-NYC (Unknown); Insight on Demand (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-088
Record Dates: First submitted 2019-02-13; First posted 2019-02-22 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Overweight; Obesity
Keywords: Focus Groups; 15-088
MeSH Terms: conditions — Overweight; Obesity | interventions — Weights and Measures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Consumo de Opciones Mas Ideales De Alimento (COMIDA) (Experimental): Participants will be placed in either individual or group interventions by convenience. Recruitment will be consecutive and participants will be placed in either intervention depending on what resource is available on a given day at the VDS, individual counselor or a group educator.
  Interventions: Behavioral: Initial in-person individual diet and exercise counseling (N vs. Y); Behavioral: Thrice weekly diet and exercise text messages (N vs. Y); Behavioral: Weekly telephone support (N vs. Y); Behavioral: Self-monitoring tools (N vs. Y) (for diet and weight)
- SANOS (Experimental): Conducting SANOS Focus Groups. We will conduct 3-5 focus groups (in Spanish) with 6-10 participants each, until saturation. Bilingual study staff will approach individuals visiting the VDS and VDS Mobile for potential participation. A brief screening questionnaire will be administered, and a BMI assessment conducted, to ascertain eligibility. Focus groups will be scheduled at the VDS Mobile unit at times convenient to participants. Participants will be verbally consented in Spanish, and will be apprised that their participation is purely voluntary and that their names will not be included in the final narrative. The 6-month follow-up and my plate dietary surveys can be done over phone. Study staff will access step counts (or obtain it through phone via the pedometer manual provided to the participant) and upload data onto the REDCap tracking tool. Staff may ask participants to report step counts captured by their personal devices (i.e., phone or smartwatch).
  Interventions: Behavioral: Initial in-person individual diet and exercise counseling (N vs. Y); Behavioral: Thrice weekly diet and exercise text messages (N vs. Y); Behavioral: Weekly telephone support (N vs. Y); Behavioral: Self-monitoring tools (N vs. Y) (for diet and weight)
- ROADmAP schema (Experimental): Participants will be randomly assigned to one of eight study groups which will be one or a combination of 4 conditions: (1) in person individualized diet and exercise counseling (2) diet and exercise text messages (3) weekly telephone support and (4) self-monitoring tools for diet and weight. For the first part of the study, Survey, approximately 64 drivers and 36 management staff will take pate in the feedback questionnaire. For the second part of the study, Interview, approximately 8 drivers and 12 management staff may be invited to take part in an interview via phone, in person, or teleconference (Zoom).
  Interventions: Behavioral: Initial in-person individual diet and exercise counseling (N vs. Y); Behavioral: Thrice weekly diet and exercise text messages (N vs. Y); Behavioral: Weekly telephone support (N vs. Y); Behavioral: Self-monitoring tools (N vs. Y) (for diet and weight)

INTERVENTIONS:
Behavioral: Initial in-person individual diet and exercise counseling (N vs. Y) — Individual counseling utilizing MI has been effective in promoting behavioral change.18 A SANOS interventionist (MRNY promotora) will deliver a 45-60 minute counseling session, utilizing MI techniques, on diet and exercise, and how to stretch one's food dollars (see description of 10 modules described above under COMIDA Pilot). The promotora will evaluate the participant's diet based on the 24-hour dietary recall132 conducted at intake (see below), will compare diet composition to the USDA's MyPlate guidelines, and will then personalize education to address identiﬁed knowledge gaps and unhealthy food choices. Promotoras will focus on goal-setting, problem solving, selfeﬃcacy enhancements, selfmonitoring skills (i.e., participants will be taught how to monitor their diet, weight, and physical activity (PA), with simple pencil-and-paper logs or with 'Self-monitoring tools' if randomized to also receive that component), and modeling of healthy behaviors.
Behavioral: Thrice weekly diet and exercise text messages (N vs. Y) — Text message interventions have been demonstrated to be effective in increasing self-eﬃcacy, weight loss, and PA.65-67 Participants will receive thrice weekly healthy eating, PA, and health care access text message tips. Links to additional information and videos will also be sent via text (e.g. local farmers markets, healthy recipes, free exercise classes, workout videos, video demonstrations of how to prepare healthy meals, etc.). Texts were developed and piloted in the COMIDA Pilot, are designed to promote goal-setting, problem-solving, self-monitoring, modeling, and self-eﬃcacy, and will be further reﬁned during the formative research phase (see below). Texts will be sent via Mosio Text Messaging Solutions. Messages will be concise, as longer messages have shown no demonstrable impact. Based on each participant's status at intake, tailored text messages will also encourage regular follow-up with PCPs. Text messages will be interactive.
Behavioral: Weekly telephone support (N vs. Y) — Several lifestyle interventions including Hispanics have successfully incorporated telephone support.134-138 Weekly telephone support (or more frequently if requested) will be delivered by the promotoras throughout the 6-month intervention. Frequent and prolonged contact in behavioral interventions is more effective than single sessions; most interventions leading to diet or PA changes persisting for >12 months have follow-up contact sessions for at least 4 months.18 Greater numbers of follow-up sessions facilitate success of behavior change, and initial behavior change can decrease with decreased contact.18,139 Telephone sessions (10-15 minutes) will use MI principles, will focus on goal-setting, problem solving, reviewing/integrating new diet/PA knowledge/skills (including self-monitoring) into individuals' daily routines, self-eﬃcacy enhancements, encouraging participants to seek opportunities for modeling and encouraging regular follow-up with PCPs.
Behavioral: Self-monitoring tools (N vs. Y) (for diet and weight) — Self-monitoring is an important component in achieving behavioral change.18 Participants will be given a SANOS food diary (adapted for and pilot-tested at the VDS in our pilot work) and a digital scale. As part of VDS Mobile usual care, all participants will receive a pedometer to assess exercise behavior (secondary outcome), so additional self-monitoring tools for PA will not be included in this component.

SUMMARY:
The Mexican Consulate runs a Ventanilla de Salud (VDS) (Health Window) program in fifty locations nationwide. The VDS provides an opportunity to provide health services to members of the Mexican community. Some of the concerns previously identified during the work at the VDS were that some individuals did not always get enough to eat, or do not always have enough money for food. This sometimes leads to unhealthy food choices-- buying and preparing foods that are inexpensive but really not good for the particpant. The investigators would like to conduct focus group to help make changes to a new diet and exercise program at the VDS called SANOS which stands for SAlud y Nutrición para todOS. SANOS aims to provide information for living a healthier lifestyle including on how to eat healthy on a small budget and how to become more physically active. The hope is that learning to eat healthy without spending a lot of money and to find simple ways to increase physical activity (like walking) will be a first step in reducing obesity rates within the Mexican community that have led to increased risks for cancer, cardiovascular disease, and diabetes.

Participants who reached 6-month follow-up during the COVID-19 pandemic, may be outside of the 12-month window post 6-month follow-up, and have not been able to complete HgbA1c and cholesterol measures will be invited to complete these measures in person at the VDS.

ELIGIBILITY:
Inclusion Criteria:

For COMIDA participants only:

* Self-Identifies as Mexican American or Mexican
* Seeking services at the VDS of the Mexican Consulate
* Prefers to speak in Spanish
* All adults at least 18 years of age
* Screens as obese (an adult who has a Body Mass Index (BMI) 30 or higher) or overweight (an adult who has a BMI between 25 - 29.9)
* Agrees to be audio recorded

For SANOS focus group participants only:

* Self-identifies as Hispanic/Latino;
* Seeking services at VDS or VDS Mobile;
* Prefers to speak in Spanish;
* At least 18 years of age;
* Screens as obese (BMI ≥ 30 kg/m^2) or overweight (BMI of 25 - 29.9 kg/m^2);
* Agrees to be audio recorded

For SANOS RCT participants only:

* Self-identifies as Hispanic/Latino;
* Seeking services at VDS or VDS Mobile;
* Prefers to speak in Spanish;
* At least 18 years of age;
* Screens as obese (BMI ≥ 30 kg/m^2) or overweight (BMI of 25 - 29.9 kg/m^2);
* Owns a cell phone capable of receiving text messages;
* Agrees to be audio recorded

For Family COMIDA participants only:

* Self-Identifies as Hispanic/Latino
* Seeking services at the VDS (or has used VDS services in the past) of the Mexican Consulate or VDS Mobile
* Prefers to speak in Spanish
* At least 18 years of age
* Has at least one child under age 18 living in the same household
* Owns a cell phone capable of receiving text messages
* Willing to receive text messages (3 texts per week for 3 months)
* Owns an internet connected device (eg, cell phone, tablet, etc) capable of conducting teleconference calls (eg, Zoom)

For ROADmAP RCT participants only:

* At least 21 years of age
* Full-time (drives at least 35 hours per week) licensed taxi/FHV driver
* Driver for at least 6 months
* Seeking Health Fairs (or has used Health Fairs services in the past)
* Speaks English, French, Bengali, or Spanish
* Screens a as obese (BMI ≥ 30 kg/m2 [≥25 kg/m2 for South Asians]) or overweight (BMI of 25 - 29.9 kg/m2 s [23- 24.9 kg/m2 for South Asians])

  * (BMI cut-offs are lower for South Asians, per WHO and American Diabetes Association recommendations)
* Owns a cell phone capable of receiving text messages
* Agrees to be audio-recorded

For ROADmAP Phase 2 participants only:

* At least 21 years of age
* Driver who participated in ROADmAP RCT or manager at a taxi garage, Uber, Lyft or driver serving/union/organization
* Agrees to be audio-recorded

Exclusion Criteria:

For COMIDA participants only:

* Will not be in the NYC area for the study duration (3-4 months) Is pregnant or might be pregnant
* Lactating women
* Presence of a chronic disease such as cancer, kidney disease, liver disease, etc. (Individuals with diabetes, lactose intolerance, and high blood pressure MAY still participate in the study)
* Has dietary restrictions (i.e. liquid diet)
* Does not have a phone that accepts text messages or unwilling to accept text messages
* Presence of a serious psychiatric or cognitive impairment likely to preclude meaningful informed consent and adherence to the protocol per the consenting professional"s judgment
* Has another family member already enrolled in COMIDA (as determined by patient report)

For SANOS focus group participants only:

* Is pregnant or might be pregnant; lactating women;
* Self-reported presence of a chronic disease such as cancer, kidney disease, liver disease, etc. (individuals with HTN and DM may still participate);
* Has dietary restrictions (i.e. liquid diet);
* Has a household member who has already participated (or agreed to participate);

For SANOS RCT participants only:

* Is pregnant or might be pregnant; lactating women; for the study duration (6 months)
* Self-reported presence of a chronic disease such as cancer, kidney disease, liver disease, etc. (individuals with HTN and DM may still participate); restricting diet;
* Currently has dietary restrictions (i.e. liquid diet);
* Has a household member who has already participated (or agreed to participate);
* Has already participated in the study
* Will not be in the NY Metropolitan area for the study duration (6 months) Works for or with the Mexican consulate (including employment and/or collaborative or volunteer services)

For Family COMIDA participants only:

* Is pregnant or might be pregnant; lactating women for the study duration (3 months)
* Will not be in the NY Metropolitan area for the study duration (3 months) Presence of a chronic disease such as cancer, kidney disease, liver disease, etc. (Individuals with diabetes, lactose intolerance, and high blood pressure MAY still participate in the study)
* Has dietary restrictions (i.e. liquid diet)
* Has another family member who has already participated in COMIDA or SANOS
* Has already participated in the study
* Works for or with the Mexican consulate (including employment and/or collaborative or volunteer services)

For ROADmAP RCT participants only:

* Is pregnant or might be pregnant; lactating women; for the study duration (12 months)
* Self-reported presence of a chronic disease such as cancer, kidney disease, liver disease, etc. (individuals with HTN and DM may still participate) that may restrict diet
* Currently has dietary restrictions (i.e. liquid diet)
* Has a household member who has already participated (or agreed to participate)
* Has already participated in the study
* Will not be in the NY Metropolitan area for 6 months from study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1785 (Estimated)
Dates: Start 2015-05-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
self-reported measures on dietary intake | 1 year
  Using the Dietary Screener of the 2011-12 California Health Interview Survey (CHIS)65 to measure diet behaviors of all participants. The information is collected through questions in the following format: "During the past month ["or in the past 7 days" for fast-food consumption], how often did you eat [food item name]?" The questions are often followed by clarification of the food items. The response is standardized to reflect mean per-week intake frequency. (Administration time ~ 10 minutes).
Decreasing weight by 5% [SANOS] | At 6 months post-intake

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Leng, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Mexican Consulate's Ventanilla de Salud (VDS), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm